CLINICAL TRIAL: NCT02931513
Title: Macrophage Activation Marker sCD163 in PBC Patients - Assessment of Treatment Response to UDCA
Brief Title: sCD163 in PBC Patients - Assessment of Treatment Response
Status: Recruiting | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: PBC AU 2
Record Dates: First submitted 2016-10-11; First posted 2016-10-13 (Estimated); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Primary Biliary Cirrhosis; Liver Inflammation; Ursodeoxycholic Acid
MeSH Terms: conditions — Liver Cirrhosis, Biliary; Hepatitis | interventions — Blood Specimen Collection; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Liverbiopsies if obtained during prognostication Blood samples for measuring sCD163 and sMR
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PBC patients: Patients with primary biliary cholangitis
  Interventions: Other: Blood samples; Device: Fibroscan; Other: Questionnaires; Biological: Liver biopsy

INTERVENTIONS:
Other: Blood samples
Device: Fibroscan
Other: Questionnaires
Biological: Liver biopsy — Liver biopsy will only be obtained if obtained as part of the diagnosis (will not be obtained for study purpose only)

SUMMARY:
Primary biliary cholangitis (PBC) is an autoimmune chronic liver disease, characterised by destruction of the small intrahepatic bile ducts. Ursodeoxycholic acid (UDCA) is the first line treatment for patients with PBC. However, up to 40% of patients respond inadequate to this treatment.

sCD163 is a macrophage activation marker shedded into plasma by macrophages in the liver. sMR is a soluble mannose receptor. The investigators want to investigate whether sCD163 and sMR can predict response to treatment with UDCA in newly diagnosed patients with PBC.

DETAILED DESCRIPTION:
Primary biliary cholangitis (PBC, previously called 'primary biliary cirrhosis') is an autoimmune cholestatic liver disease characterized by destruction of intrahepatic bile ducts and progression to liver fibrosis and cirrhosis. In the pre-cirrhotic phase, fatigue and pruritus are the dominant symptoms. These symptoms reduce PBC patients' quality of life, but the extent to which they cause the patient to leave the work force and seek disability pension is unknown. The diagnosis of PBC is based on the presence of two of three major criteria; unexplained serum alkaline phosphatase (ALP) >1.5 times upper normal limit for more than 24 weeks, presence of anti-mitochondrial antibodies (AMA), and compatible liver histology. Multiple models have been conducted to predict prognosis in patients with PBC. The Mayo risk score is the best validated and includes information on age, bilirubin, albumin, prothrombin time and peripheral oedema. Other prognostic factors are pruritus and fatigue at diagnosis that predict the time to develop cirrhosis and its complications.

Ursodeoxycholic acid is the first line treatment for all patients with PBC. Response to treatment is assessed after 12 months of treatment using e.g. the Paris 1 criteria (ALP <3 times upper normal limit, AST <2 times upper normal limit, and bilirubin ≤1 mg/dL after one year of treatment). Up to 40% of patients respond inadequately to UDCA and need add-on therapies. (e.g. fibrates, budenosid or obeticholic acid).

In PBC, inflammation is attributed to an immune response to mitochondrial autoantigens followed by a serologic response of anti-mitochondrial antibodies (AMAs); and accompanied by inflammation of small bile ducts. The pathogenesis includes both CD4 and CD8 cells, which in the presence of biliary cells expressing the 2-oxo-dehydrogenase pathway (PDC-E2) activates macrophages via granulocyte macrophage colony-stimulating factor. The activated macrophages, together with AMAs, produce a proinflammatory response with subsequent liver inflammation and fibrosis. Thus, macrophages seem to be involved in PBC disease severity and progression. However, macrophage activation markers have not previously been investigated in PBC patients. The investigators in our research group have during the last years investigated the macrophage activation marker sCD163. The group have shown increased levels in relation to liver fibrosis/cirrhosis in patients with chronic viral hepatitis (HBV and HCV), non-alcoholic fatty liver disease (NAFLD/NASH) and alcoholic liver disease (alcoholic hepatitis and cirrhosis) and liver disease severity including risk of portal hypertension and development of complications and mortality. Just recently the investigators' group also demonstrated that the soluble mannose receptor (sMR) and sCD163 are associated with early and long-term prognosis of patients with cirrhosis and acute-on-chronic liver failure.

Aims:

To investigate sCD163 and sMR at diagnosis, before treatment with UDCA, as possible predictors of non-response to UDCA treatment and thus as predictors of patients needing add-on therapy.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed with Primary biliary cholangitis
* No treatment with UDCA

Exclusion Criteria:

* Patient under 18 years
* Expected lifetime under 6 months
* Expected liver transplantation within 6 months
* Liver cancer
* Cirrhosis from other causes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with primary biliary cholangitis seen at Aarhus University Hospital, Aarhus, Denmark or at any regional hospital in the Central Region of Denmark
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2016-09; Primary Completion 2031-01 (Estimated); Study Completion 2031-09 (Estimated)

PRIMARY OUTCOMES:
UDCA response (ALP <3 times upper normal limit, AST <2 times upper normal limit, and bilirubin ≤1 mg/dL after one year of treatment) | 1 year

SECONDARY OUTCOMES:
disease progression (blood samples, fibroscan, questionnaires) | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Hepatology and Gastroenterology, Aarhus University Hospital, Denmark, Aarhus C, Central Jutland, Denmark

IPD SHARING:
Plan to Share IPD: Undecided